CLINICAL TRIAL: NCT00685919
Title: Kidney Dopamine Effects on Urinary Sodium Excretion in Postural Tachycardia Syndrome
Brief Title: Peripheral Dopamine in Postural Tachycardia Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alfredo Gamboa, Research Associate Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 101499; HL071784-05A1
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Postural Tachycardia Syndrome; Orthostatic Intolerance
Keywords: Dopamine; Natriuresis; Catecholamines
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance | interventions — Carbidopa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbidopa then Placebo (Experimental): Carbidopa 200 mg every 6 hours orally for 5 doses followed by Placebo every 6 hours for 5 doses
  Interventions: Drug: Carbidopa; Drug: Placebo
- Placebo then Carbidopa (Experimental): Placebo matching carbidopa given every 6 hours orally for 5 doses followed by Carbidopa
  Interventions: Drug: Carbidopa; Drug: Placebo

INTERVENTIONS:
Drug: Carbidopa — 200 mg every 6 hours for 5 doses given orally
Drug: Placebo — every 6 hours for 5 doses, given orally, and matching Carbidopa

SUMMARY:
The purpose of the proposed research is to determine how changes in kidney dopamine (DA) activity influence urinary sodium excretion. We will decrease DA activity in the kidney by inhibiting DA synthesis via carbidopa administration. We want to compare findings in normal volunteers and in patients with postural tachycardia syndrome (POTS). We will test the null hypothesis (Ho) that the effects of oral carbidopa administration on urinary sodium excretion will not differ between patients with POTS and healthy volunteers.

DETAILED DESCRIPTION:
We will determine whether inhibition of renal dopamine formation by carbidopa administration leads to a decrease in urinary excretion of dopamine and sodium and whether the response differs in POTS and control populations. Carbidopa effects will be compared to those of a matching placebo, and the sequence of treatments (carbidopa before placebo or placebo before carbidopa) will be randomized.

Each subject will undergo a complete history and physical examination, including an electrocardiogram (EKG).

* After achieving sodium balance on a 200 mEq/day sodium diet, subjects will collect urine over 24hr for baseline assessment of sodium and catecholamines.
* On this day, the subjects will be admitted to the CRC.
* An 18 gauge intravenous catheter will be inserted in order to draw blood.
* The subjects will fast from 7 pm until after the next morning's testing.
* In the morning, while still supine after the overnight sleep, heart rate and blood pressure will be recorded, and blood will be drawn. The subjects will then stand for 10 minutes. Heart rate and blood pressure will be measured at intervals, and an upright blood sample will be collected.
* The subjects will be asked to collect their urine to end the 24hr urine collection. Another 24hr urine collection will be started.
* Treatment A (Carbidopa 200mg or placebo) will be given orally following the void, at approximately 7 am. Additional doses will be taken every 6 hours with the last dose at 7 am the following morning.
* Subjects will be free to follow their normal routine during the day until returning to the CRC for the night. However, they will need to consume the 200 mEq/day study diet for each meal, collect all urine, and take study medication on schedule
* After returning to the CRC, the subjects will fast after 7 pm.
* In the morning, supine and standing heart rate and blood pressure will be recorded, and the subjects will be asked to collect their urine to end the 24hr urine collection.
* The final dose of study medication (Carbidopa 200mg or placebo) will be given orally following the void, at approximately 7 am.
* Supine heart rate and blood pressure will be measured and supine blood samples will be collected hourly for 4 hours after the treatment and at 8 hours after the treatment. Subjects must rest supine for at least 30 minutes before each blood draw.
* At 2 hours after treatment, subjects will stand for 10 minutes for upright blood pressure and heart rate measurements and collection of an upright blood sample, as described above. Participants will be asked to rate the severity of common orthostatic symptoms while supine and upright.
* Urine will be collected for two 4-hour periods after treatment and from 8 hours to 24 hours after treatment.
* Fixed-sodium study diet will be provided after the 4-hour measurements and in the evening.

After at least a 1 day washout period, the study will be repeated with Treatment B

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with POTS by the Vanderbilt Autonomic Dysfunction Center based on the following stringent criteria: 1) history of daily orthostatic symptoms for at least 6 months; 2) increase in heart rate (HR) of at least 30 bpm with standing or a standing HR of at least 120 bpm; 3) absence of orthostatic hypotension (defined as a fall in blood pressure (BP)>20/10 mm Hg); and 4) absence of conditions, such as dehydration, substantial weight loss, or systemic illnesses, that could provoke orthostatic intolerance
* Upright plasma NE at least 600 pg/mL in patients
* Non-smoking
* Free of medications with the potential to influence BP
* Able and willing to provide informed consent -

Exclusion Criteria:

* Overt cause for postural tachycardia (such as acute dehydration)
* Significant cardiovascular, pulmonary, hepatic, or hematological disease by history or screening results
* Positive urine b-hcg pregnancy test
* Evidence of cardiac structural disease (by clinical examination or prior echocardiogram)
* Hypertension defined as a BP>145/95 (off medications) or need for antihypertensive medications
* Evidence of significant conduction system delay (QRS duration >120 ms) on electrocardiogram
* Inability to give, or withdraw, informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo J Gamboa, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Carey RM. Theodore Cooper Lecture: Renal dopamine system: paracrine regulator of sodium homeostasis and blood pressure. Hypertension. 2001 Sep;38(3):297-302. doi: 10.1161/hy0901.096422. PMID 11566894
- [Background] Goldstein DS, Stull R, Eisenhofer G, Gill JR Jr. Urinary excretion of dihydroxyphenylalanine and dopamine during alterations of dietary salt intake in humans. Clin Sci (Lond). 1989 May;76(5):517-22. doi: 10.1042/cs0760517. PMID 2498027
- [Background] Jose PA, Eisner GM, Felder RA. Renal dopamine and sodium homeostasis. Curr Hypertens Rep. 2000 Apr;2(2):174-83. doi: 10.1007/s11906-000-0079-y. PMID 10981146
- [Background] Kuchel O, Buu NT, Unger T. Dopamine-sodium relationship: is dopamine a part of the endogenous natriuretic system? Contrib Nephrol. 1978;13:27-36. doi: 10.1159/000402132. PMID 710137
- [Background] Stokes GS, Monaghan JC, Pillai DN. Effects of carbidopa and of intravenous saline infusion into normal and hypertensive subjects on urinary free and conjugated dopamine. J Hypertens. 1997 Jul;15(7):761-8. doi: 10.1097/00004872-199715070-00008. PMID 9222944
- [Background] Jacob G, Robertson D, Mosqueda-Garcia R, Ertl AC, Robertson RM, Biaggioni I. Hypovolemia in syncope and orthostatic intolerance role of the renin-angiotensin system. Am J Med. 1997 Aug;103(2):128-33. doi: 10.1016/s0002-9343(97)00133-2. PMID 9274896

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: * Healthy Participants Group: 21 healthy controls enrolled. 3 withdrew prior to randomization. 1 screen failed. 17 healthy participants were randomized. 1 participant was withdrawn due to orthostatic symptoms during baseline testing
  * Postural Tachycardia Syndrome (POTS) Group: 11 POTS participants were randomized. 1 participant withdrew after the 1st dose of the intervention (placebo).
Groups:
- Healthy Participants-Placebo Then Carbidopa; Patients With POTS-Placebo Then Carbidopa: Placebo every 6 hours for 5 doses followed by Carbidopa 200 mg every 6 hours orally for 5 doses
- Healthy Participants-Carbidopa Then Placebo; Patients With POTS-Carbidopa Then Placebo: Carbidopa 200 mg every 6 hours for 5 doses followed by Placebo given orally every 6 hours for 5 doses
Period: Overall Study
Arm/Group | Healthy Participants-Placebo Then Carbidopa | Healthy Participants-Carbidopa Then Placebo | Patients With POTS-Placebo Then Carbidopa | Patients With POTS-Carbidopa Then Placebo
Started | 8 (8 healthy controls were randomized to receive placebo followed by carbidopa. 1 received only 50 mg doses of carbidopa and her data were excluded.) | 9 (9 healthy controls were randomized to receive carbidopa followed by placebo.) | 8 (8 patients with POTS were randomized to receive placebo followed by carbidopa. 1 of these received only 50 mg doses of carbidopa and her data are excluded.) | 3 (3 patients with POTS were randomized to receive carbidopa followed by placebo.)
Baseline A | 8 (After achieving sodium balance on 200 mEq/day sodium diet, subjects collected baseline 24hr urine. They fasted from 7pm until the next morning. In the morning, while still supine, heart rate and blood pressure were recorded and blood was drawn. Participants then stood for 10 min. Heart rate and blood pressure were measured at intervals and an upright blood sample was collected. Urine was collected to end the 24hr collection.) | 9 (After achieving sodium balance on 200 mEq/day sodium diet, subjects collected baseline 24hr urine. They fasted from 7pm until the next morning. In the morning, while still supine, heart rate and blood pressure were recorded and blood was drawn. Participants then stood for 10 min. Heart rate and blood pressure were measured at intervals and an upright blood sample was collected. Urine was collected to end the 24hr collection. 1 patient withdrew after orthostatic symptoms during baseline.) | 8 (After achieving sodium balance on 200 mEq/day sodium diet, subjects collected baseline 24hr urine. They fasted from 7pm until the next morning. In the morning, while still supine, heart rate and blood pressure were recorded and blood was drawn. Participants then stood for 10 min. Heart rate and blood pressure were measured at intervals and an upright blood sample was collected. Urine was collected to end the 24hr collection. 1 patient withdrew after orthostatic symptoms during baseline.) | 3 (After achieving sodium balance on 200 mEq/day sodium diet, subjects collected baseline 24hr urine. They fasted from 7pm until the next morning. In the morning, while still supine, heart rate and blood pressure were recorded and blood was drawn. Participants then stood for 10 min. Heart rate and blood pressure were measured at intervals and an upright blood sample was collected. Urine was collected to end the 24hr collection.)
Treatment A | 7 (Following the urine collection to end the baseline urine and the baseline testing, placebo was given orally. Additional doses were given every 6 hours with the last dose at 7am the following morning. Urine was collected over 24hr and supine and upright heart rates, blood pressures and blood samples were collected.) | 9 (Following the urine collection to end the baseline urine and the baseline testing, carbidopa 200 mg was given orally. Additional doses were given every 6 hours with the last dose at 7am the following morning. Urine was collected over 24hr and supine and upright heart rates, blood pressures and blood samples were collected.) | 8 (Following the urine collection to end the baseline urine and the baseline testing, placebo was given orally. Additional doses were given every 6 hours with the last dose at 7am the following morning. Urine was collected over 24hr and supine and upright heart rates, blood pressures and blood samples were collected.) | 3 (Following the urine collection to end the baseline urine and the baseline testing, carbidopa 200 mg was given orally. Additional doses were given every 6 hours with the last dose at 7am the following morning. Urine was collected over 24hr and supine and upright heart rates, blood pressures and blood samples were collected.)
24 hr Post-treatment A | 7 (Urine was collected for 24 hr after the last dose of Treatment A.) | 9 (Urine was collected for 24 hr after the last dose of Treatment A.) | 7 (Urine was collected for 24 hr after the last dose of Treatment A.) | 3 (Urine was collected for 24 hr after the last dose of Treatment A.)
Baseline B | 7 (After at least a 1-day washout period, patients underwent baseline procedures as described previously.) | 9 (After at least a 1-day washout period, patients underwent baseline procedures as described previously.) | 7 (After at least a 1-day washout period, patients underwent baseline procedures as described previously.) | 3 (After at least a 1-day washout period, patients underwent baseline procedures as described previously.)
Treatment B | 7 (Following the urine collection to end the baseline urine and the baseline testing, carbidopa 200 mg was given orally. Additional doses were given every 6 hours with the last dose at 7am the following morning. Urine was collected over 24hr and supine and upright heart rates, blood pressures and blood samples were collected.) | 9 (Following the urine collection to end the baseline urine and the baseline testing, placebo was given orally. Additional doses were given every 6 hours with the last dose at 7am the following morning. Urine was collected over 24hr and supine and upright heart rates, blood pressures and blood samples were collected.) | 7 (Following the urine collection to end the baseline urine and the baseline testing, carbidopa 200 mg was given orally. Additional doses were given every 6 hours with the last dose at 7am the following morning. Urine was collected over 24hr and supine and upright heart rates, blood pressures and blood samples were collected.) | 3 (Following the urine collection to end the baseline urine and the baseline testing, placebo was given orally. Additional doses were given every 6 hours with the last dose at 7am the following morning. Urine was collected over 24hr and supine and upright heart rates, blood pressures and blood samples were collected.)
24 hr Post Treatment B | 7 (Urine was collected for 24 hr after last dose of Treatment B.) | 9 (Urine was collected for 24 hr after last dose of Treatment B.) | 7 (Urine was collected for 24 hr after last dose of Treatment B.) | 3 (Urine was collected for 24 hr after last dose of Treatment B.)
Completed | 7 | 9 | 7 | 3
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: * Healthy Participant Group: Data is excluded for 1 participant who was withdrawn due to orthostatic symptoms during baseline testing.
  * Postural Tachycardia Syndrome (POTS) Group: Data is excluded for 1 participant who was withdrawn after the 1st dose of the intervention (placebo).
Groups:
- POTS-Carbidopa Then Placebo: Carbidopa 200 mg every 6 hours for 5 doses followed by Placebo given orally every 6 hours for 5 doses
- Total: Total of all reporting groups
Arm/Group | Healthy Participants-Placebo Then Carbidopa | Healthy Participants-Carbidopa Then Placebo | Patients With POTS-Placebo Then Carbidopa | POTS-Carbidopa Then Placebo | Total
Number analyzed (Participants) | 8 | 8 | 7 | 3 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 32 (10) | 31 (10) | 37 (3) | 32.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 3 | 25
  Male | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 7 | 3 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 8 | 7 | 7 | 3 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 7 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Urinary Sodium Excretion During Treatment Normalized to Creatinine
Description: Urine was collected for 24hr during treatment. Urinary volume was measured and the urine was analyzed for sodium and creatinine concentrations. Total amounts of sodium and creatinine excreted over the 24 hr were calculated and results expressed as ratio of sodium:creatinine.
Time Frame: Immediately before the 1st dose of placebo or carbidopa to immediately before the 5th dose (approximately 24 hours)
Population: No data analysis for the following:
  Healthy Placebo Group:
  * 1 subject with discarded urine sample
  * 1 subject who received only 50mg carbidopa (data for all arms excluded)
  Healthy Carbidopa Group:
  * 1 subject who received only 50mg carbidopa (wrong dose)
  POTS Placebo Group:
  * 1 subject with discarded urine sample
  * 1 subject who received only 50mg carbidopa (data for all arms excluded)
  POTS Carbidopa Group:
  * 1 subject who received only 50mg carbidopa (wrong dose)
Measure: Mean (Standard Deviation); unit: Milliequivalents per gram (mEq/g)
Groups:
- Healthy Participants Who Received Placebo as Treatment A or Treatment B: Healthy participants received Placebo matching Carbidopa given every 6 hours orally for 5 doses
- Healthy Participants Who Received Carbidopa as Treatment A or Treatment B: Healthy participants received Carbidopa: 200 mg every 6 hours for 5 doses given orally
- Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B: POTS participants received Placebo matching carbidopa given every 6 hours orally for 5 doses
- Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B: POTS participants received Carbidopa: 200 mg every 6 hours for 5 doses given orally
Arm/Group | Healthy Participants Who Received Placebo as Treatment A or Treatment B | Healthy Participants Who Received Carbidopa as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B
Number analyzed (Participants) | 14 | 15 | 8 | 9
Milliequivalents per gram (mEq/g) | 140 (29) | 132 (38) | 137 (30) | 154 (31)

2. Secondary Outcome: Systolic Blood Pressure Measured at 8 Hours After the Last Dose of Placebo or Carbidopa
Description: Systolic blood pressure was measured once using a Dinamap non-invasive oscillometric blood pressure monitor, 2-4 hours after lunch and after at least 30 minutes of resting supine.
Time Frame: 8 hours after the last dose of placebo or carbidopa
Population: No data analysis for the following:
  Healthy Placebo Group:
  * 1 subject with missing systolic blood pressure 8-hours after the last dose of Placebo
  * 1 subject who received only 50mg carbidopa (data for all arms excluded)
  Healthy Carbidopa Group:
  * 1 subject who received only 50mg carbidopa (wrong dose)
  POTS Placebo Group:
  * 1 subject who received only 50mg carbidopa (data for all arms excluded)
  POTS Carbidopa Group:
  * 1 subject who received only 50mg carbidopa (wrong dose)
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Healthy Participants Who Received Placebo as Treatment A or Treatment B | Healthy Participants Who Received Carbidopa as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B
Number analyzed (Participants) | 14 | 15 | 9 | 9
millimeters of mercury (mmHg) | 103 (4) | 101 (8) | 102 (9) | 101 (10)

3. Secondary Outcome: Plasma Catecholamines (Norepinephrine) After the Last Dose of Placebo or Carbidopa
Description: Blood samples were collected while resting supine for at least 30 minutes and 2 to 4 hours after lunch. For catecholamine measurements, blood was collected in chilled vacuum tubes with EDTA. Plasma was separated and stored with added reduced glutathione (Amersham International PLC) at -70°C until the assay. Plasma catecholamines were measured by a method that involves batch alumina extraction followed by high-performance liquid chromatography (HPLC) for separation with electrochemical detection and quantification.
Time Frame: 8 hours after the last dose of placebo or carbidopa
Population: No data analysis for the following:
  Healthy Placebo Group:
  * 1 subject who received only 50mg carbidopa (data for all arms excluded)
  Healthy Carbidopa Group:
  * 1 subject who received only 50mg carbidopa (wrong dose)
  POTS Placebo Group:
  * 1 subject who received only 50mg carbidopa (data for all arms excluded)
  POTS Carbidopa Group:
  * 1 subject who received only 50mg carbidopa (wrong dose)
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Healthy Participants Who Received Placebo as Treatment A or Treatment B | Healthy Participants Who Received Carbidopa as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B
Number analyzed (Participants) | 15 | 15 | 9 | 9
Picograms per milliliter (pg/mL) | 150 (46) | 181 (100) | 278 (84) | 245 (70)

4. Secondary Outcome: Plasma Catecholamines (DOPA) After the Last Dose of Placebo or Carbidopa
Description: as for outcome 3
Time Frame: 8 hours after the last dose of placebo or carbidopa
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Healthy Participants Who Received Placebo as Treatment A or Treatment B | Healthy Participants Who Received Carbidopa as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B
Number analyzed (Participants) | 15 | 15 | 9 | 9
Picograms per milliliter (pg/mL) | 1813 (463) | 20297 (9509) | 2104 (700) | 25680 (13825)

5. Secondary Outcome: 24 Hour Urinary Catecholamine (DOPA) Excretion During Treatment Normalized to Creatinine
Description: Urine was collected over 24 hours during treatment. The urinary volume was measured and the urine was analyzed for creatinine and catecholamines. Total amounts of creatinine and catecholamines were calculated and the results are expressed as catecholamine:creatinine.
Time Frame: Immediately before the 1st dose of Placebo or Carbidopa and ending immediately before the last dose (approximately 24 hours)
Population: No data analysis for the following participants:
  Healthy Placebo:
  * 1 w/ discarded urine sample
  * 1 w/ urine not analyzed for catecholamines
  * 1 received only 50mg carbidopa (data for all arms excluded)
  Healthy Carbidopa:
  * 1 w/ urine not analyzed for catecholamines
  * 1 received only 50mg carbidopa (wrong dose)
  POTS Placebo:
  * 1 w/ discarded urine sample
  * 1 received only 50mg carbidopa (data for all arms excluded)
  POTS Carbidopa:
  * 1 received only 50mg carbidopa (wrong dose)
Measure: Mean (Standard Deviation); unit: Micrograms per milligrams (ug/mg)
Arm/Group | Healthy Participants Who Received Placebo as Treatment A or Treatment B | Healthy Participants Who Received Carbidopa as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B
Number analyzed (Participants) | 13 | 14 | 8 | 9
Micrograms per milligrams (ug/mg) | 0.024 (0.014) | 0.283 (0.194) | 0.026 (0.015) | 0.385 (0.156)

6. Secondary Outcome: 24 Hour Urinary Catecholamine (Dopamine) Excretion During Treatment Normalized to Creatinine
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Micrograms per milligrams (ug/mg)
Arm/Group | Healthy Participants Who Received Placebo as Treatment A or Treatment B | Healthy Participants Who Received Carbidopa as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B
Number analyzed (Participants) | 13 | 14 | 8 | 9
Micrograms per milligrams (ug/mg) | 0.208 (0.061) | 0.035 (0.015) | 0.24 (0.081) | 0.038 (0.015)

7. Secondary Outcome: Supine Plasma Renin Activity 2 Hours After the Last Dose of Placebo or Carbidopa
Description: Blood samples were collected while resting supine for at least 30 minutes and 1 1/2 to 2 hours after breakfast. Samples were processed and sent to the Vanderbilt Clinic Laboratory for assay.
Time Frame: 2 hours after the last dose of placebo or carbidopa
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter per hour (ng/mL
Arm/Group | Healthy Participants Who Received Placebo as Treatment A or Treatment B | Healthy Participants Who Received Carbidopa as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B
Number analyzed (Participants) | 15 | 15 | 9 | 9
Nanograms per milliliter per hour (ng/mL | 1.153 (0.926) | 1.033 (0.529) | 1.544 (1.02) | 1.878 (1)

8. Secondary Outcome: Plasma Sodium After the Last Dose of Placebo or Carbidopa
Description: Blood samples were collected while resting supine for at least 30 minutes and 2 to 4 hours after lunch. Samples were processed and sent to the Vanderbilt Clinical Laboratory for assay.
Time Frame: 8 hours after the last dose of placebo or carbidopa
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliequivalents per liter (mEq/L)
Arm/Group | Healthy Participants Who Received Placebo as Treatment A or Treatment B | Healthy Participants Who Received Carbidopa as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Participants Who Received Placebo as Treatment A or Treatment B | Postural Tachycardia Syndrome (POTS) Patients Who Received Carbidopa as Treatment A or Treatment B
Number analyzed (Participants) | 15 | 15 | 9 | 9
Milliequivalents per liter (mEq/L) | 138 (1.9) | 138 (1.9) | 139 (2.2) | 138 (2)

ADVERSE EVENTS:
Time Frame: Participants were followed for 24 hours after the 5th dose of treatment.
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Events were self-reported by participants.
Groups:
- Healthy Participants-Placebo; POTS Participants-Placebo: Placebo matching carbidopa given every 6 hours orally for 5 doses
- Healthy Participants-Carbidopa; POTS Participants-Carbidopa: Carbidopa 200 mg every 6 hours orally for 5 doses
Arm/Group | Healthy Participants-Placebo | Healthy Participants-Carbidopa | POTS Participants-Placebo | POTS Participants-Carbidopa
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/17 | 1/17 | 2/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants-Placebo (N=17) | Healthy Participants-Carbidopa (N=17) | POTS Participants-Placebo (N=11) | POTS Participants-Carbidopa (N=11)
Head rush (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-04-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT00685919/Prot_SAP_ICF_000.pdf